CLINICAL TRIAL: NCT05506787
Title: Effects of Intraoperative Low-dose S-ketamine on Postoperative Mood and Pain in Patients With Crohn's Disease Undergoing Enterectomy With Mild to Moderate Depression: a Randomized Controlled Trial
Brief Title: The Effects of Intraoperative Esketamine on Postoperative Pain and Mood in Patients With Inflammatory Bowel Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Zhang Zhen, resident doctor, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2020NZKY-062-01
Record Dates: First submitted 2022-08-14; First posted 2022-08-18 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Crohn Disease; Depression; Esketamine
MeSH Terms: conditions — Crohn Disease; Depression | interventions — Esketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Esketamine Group (Experimental): The patients in S-ketamine group received 0.25 mg/kg intravenous S-ketamine (Jiangsu Hengrui Pharmaceutical Co., Ltd., Jiangsu, China) drip under general anesthesia induction, followed by continuous infusion of S-ketamine with 0.12 mg/kg/h for more than 30 minutes through target-controlled infusion. Drug A: S-ketamine, diluted to 1mg/ml with normal saline, total 50ml).
  Interventions: Drug: Esketamine
- Placebo Group (Placebo Comparator): Patients in Placebo group received intravenous infusion of 0.9% saline during anesthesia induction and were maintained through the infusion pump of drug B (50 ml 0.9% saline) for more than 30 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esketamine — Esketamine
  Arms: Esketamine Group
Drug: Placebo — Placebo
  Arms: Placebo Group

SUMMARY:
Crohn's disease (CD) is a chronic inflammatory disease of the gastrointestinal tract with symptoms evolving in a relapsing and remitting manner. Typically, the peak incidence of CD is 18 to 35 years , which means that patients with CD will be plagued by the disease during their most precious years, and nearly 35% of them will develop depressive symptoms. For 70% of patients with CD who need surgery, the incidence of preoperative depression may be higher. The CD cohort with diagnosable psychological condition has been shown to experience a higher rate of disease exacerbation than the CD cohort without psycho complication. At the same time, this depressive mood may make postoperative recovery more difficult, so it is necessary to alleviate postoperative depression.

Ketamine, a widely used anesthetic, is also used to treat depression. The most used ketamine in clinical practice is racemic ketamine, but its use is associated with many complications such as psychotic adverse effects and neurotoxicity. In recent years, S-ketamine has received attention for better efficacy and fewer complications . In 2019, the Food and Drug Administration (FDA) approved S-ketamine nasal spray for the treatment of refractory depression and subsequently received approval from numerous health authorities around the world. This proves that S-ketamine can provide a rapid antidepressant effect in patients with depression in a non-surgical setting. However, it is inconclusive whether S-ketamine affects surgical patients, mainly because of differences in the type of surgery, the dosage administered, the interaction with analgesics, and the evaluation tools implemented. Studies have shown that small doses of S-ketamine in breast cancer surgery and cervical cancer surgery can reduce postoperative depression. However, the effects of S-ketamine on postoperative depression (POD) and pain in patients with CD have not been studied.

ELIGIBILITY:
Inclusion Criteria:

1. subjects who volunteered and signed informed consent for the trial, (b) patients aged between 18 and 60, (c) patients with CD who underwent surgery, (d) American Society of Anesthesiologists (ASA) grade Ⅰ~Ⅲ, (e) Hamilton depression score 8-24.

Exclusion Criteria:

1. allergy to narcotic drugs or ketamine used, (b) patients with other serious systemic diseases (including severe heart, kidney, and liver disease), (c) chronic opioid therapy (more than twice a week for more than three months), (d) inability to understand the digital pain scale, (e) Hamilton depression score < 8 or > 24.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
the HAMD-17 score on the 7th day postoperatively | on the 7th day postoperatively
  HAMD-17, Hamilton Depression Scale 17-item (0-54 score) The total score was more than 24 as severe depression, more than 17 as mild or moderate depression, and less than 7 as no depressive symptoms.
  The higher the total score, the higher the degree of depression

SECONDARY OUTCOMES:
the HAMD-17 score at 1 day, 3 days and 30 days postoperatively | at 1 day, 3 days and 30 days postoperatively
  HAMD-17, Hamilton Depression Scale 17-item (0-54 score) The total score was more than 24 as severe depression, more than 17 as mild or moderate depression, and less than 7 as no depressive symptoms.
  The higher the total score, the higher the degree of depression
the NRS scores at PACU, 1 day, 2 days and 7 days postoperatively | baseline (at PACU), 1 day, 2 days and 7 days postoperatively
  NRS, numeric rating scale The digital pain score scale uses 0-10 points to represent different degrees of pain, 0 for no pain and 10 for severe pain. Patients score pain according to their own subjective feelings.
  Score criteria:
  0: painless 1-3: mild pain 4-6: moderate pain 7-10: severe pain
the level of C-reactive Protein (CRP) at 1 day and 3 days postoperatively | at 1 day and 3 days postoperatively
the level of interleukin 6 (IL-6) at 1 day and 3 days postoperatively | at 1 day and 3 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Ji Qing, Study Director — Anesthesiology Department, Jinling Hospital Affiliated to Nanjing University
Locations (1):
- Anesthesiology Department, Jinling Hospital Affiliated to Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No